CLINICAL TRIAL: NCT03388749
Title: Phase 1/2 Study of Liposomal Annamycin for the Treatment of Subjects With Acute Myeloid Leukemia (AML) That is Refractory to or Relapsed After Induction Therapy
Brief Title: Study of Liposomal Annamycin for the Treatment of Subjects With Acute Myeloid Leukemia (AML)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Moleculin Biotech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MB-105
Record Dates: First submitted 2017-12-25; First posted 2018-01-03 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Leukemia, Myeloid, Acute
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Liposomal annamycin (Experimental)
  Interventions: Drug: Liposomal Annamycin

INTERVENTIONS:
Drug: Liposomal Annamycin — 2-hour intravenous infusion liposomal annamycin daily for 3 consecutive days followed by 18 days off study drug (i.e., one treatment cycle = 21 days).

SUMMARY:
This is a multi-center, open-label, dose escalation study that will determine the maximum tolerated dose (MTD) and recommended Phase 2 dose (RP2D) of liposomal annamycin as a single agent for the treatment of subjects with AML that is refractory to or relapsed after induction therapy

DETAILED DESCRIPTION:
Enrollment will occur in cohorts of 3 subjects in a conventional 3+3 escalating dose design, starting at a dose level of 120 mg/m2/day administered for 3 days. Dose escalation will take place on the basis of safety assessments in sequential cohorts of 3 subjects each. The initial cohort will receive 120 mg/m2/day for 3 days. For Cohorts 1, 2, 3, 4, and 5, dose escalation will occur in 30-mg/m2/day increments until subjects are enrolled at a 240-mg/m2/day dose. For Cohorts 6, 7, and 8, dose escalation will occur in 60-mg/m2/day increments until subjects are enrolled at a maximum dose of 420 mg/m2/day. Thus subsequent cohorts will receive 150, 180, 210, 240, 300, 360, and up to a maximum of 420 mg/m2/day for 3 days in the absence of safety concerns.

In each cohort during the dose escalation phase, if 1 of the 3 subjects experiences a DLT, the cohort of subjects at that dose level will be expanded to 6 subjects. If at least 2 of the 6 subjects experience a DLT, this will be considered a toxic dose and the next 3 subjects will be treated at a lower dose. The dose will be de-escalated in 30-mg/m2/day increments. As such, if at least 2 out of 6 subjects receiving 300, 360, or 420 mg/m2/day experience a DLT, the next 3 subjects will receive 270, 330, or 390 mg/m2/day, respectively. The MTD is defined as the highest dose of L-Annamycin at which fewer than 2 (of a cohort of up to 6) subjects experience a DLT.

Once the MTD/RP2D is identified, up to 21 additional subjects will be enrolled at the MTD/RP2D to better define toxicity and evaluate efficacy at this dose.

ELIGIBILITY:
Inclusion Criteria

1. Subjects have a pathologically confirmed diagnosis of AML by World Health Organization classification.
2. Subjects have AML that is refractory to or relapsed after induction therapy (i.e., subjects relapsed after experiencing a CR with their prior therapy). To be defined as relapse, there must be >5% blasts in the bone marrow.
3. Subjects are age ≥18 years at the time of signing informed consent.
4. Subjects have not received chemotherapy, radiation, or major surgery within 2 weeks prior to first dose of study drug and/or have recovered from the toxic side effects of any previous therapy, unless treatment is indicated as a result of progressive disease, such as hydroxyurea.
5. Subjects have not received investigational therapy within 4 weeks of the first dose of study drug.
6. Subjects have an Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2.
7. Subjects have adequate laboratory results including the following:

   1. Bilirubin ≤2 times the upper limit of normal unless due to Gilbert Syndrome or leukemic infiltration of the liver
   2. Alanine aminotransferase (serum glutamic pyruvic transaminase), aspartate aminotransferase (serum glutamic-oxaloacetic transaminase), and alkaline phosphatase <2.5 times the upper limit of normal unless due to organ involvement.
   3. Adequate renal function with creatinine levels ≤2 times the upper limit of normal.
8. Subjects can understand and sign the informed consent document, can communicate with the Investigator, and can understand and comply with the requirements of the protocol.
9. Women of childbearing potential must have a negative serum or urine pregnancy test.
10. All men and women must agree to practice effective contraception during the entire study period and after discontinuing study drug, unless documentation of infertility exists.

    1. Sexually active, fertile women must use 2 effective forms of contraception (abstinence, intrauterine device, oral contraceptive, or double barrier device) from the time of informed consent and until at least 6 months after discontinuing study drug.
    2. Sexually active men and their sexual partners must use effective contraceptive methods from the time of subject informed consent and until at least 3 months after discontinuing study drug.

Exclusion Criteria

1. Subjects have been diagnosed with acute promyelocytic leukemia.
2. The subjects are receiving concomitant therapy that includes other chemotherapy that is or may be active against AML, except agents such as hydroxyurea, used to control the WBC count until chemotherapy, up to Day 1 of L-Annamycin administration.
3. Subjects have any condition that, in the opinion of the Investigator, places the subject at unacceptable risk if they were to participate in the study.
4. Subjects have central nervous system involvement.
5. Subjects have left ventricular ejection fraction (LVEF) <50%, valvular heart disease, or severe hypertension. Cardiac subjects with a New York Heart Association classification of 3 or 4 will be excluded. (Cardiology consultation should be requested if any question arises about cardiac function.) This also includes subjects with baseline QT/QTc interval >480 msec, subjects with a history of additional risk factors for torsade des pointes (e.g., heart failure, hypokalemia, family history of Long QT Syndrome), and subjects who use concomitant medications that significantly prolong the QT/QTc interval.
6. Subjects have clinically relevant serious comorbid medical conditions including, but not limited to, active infection, recent (less than or equal to 6 months) myocardial infarction, unstable angina, symptomatic congestive heart failure, uncontrolled hypertension, uncontrolled cardiac arrhythmias, chronic obstructive or chronic restrictive pulmonary disease, known positive status for human immunodeficiency virus and/or active hepatitis B or C, cirrhosis, or psychiatric illness/social situations that would limit compliance with study requirements.
7. Subjects are pregnant, lactating, or not using adequate contraception.
8. Subjects have a known allergy to anthracyclines.
9. Subjects have ongoing Grade 1 mucositis at the time of entry.
10. Subjects are required to use moderate or strong inhibitors and inducers of Cytochrome P450 family of enzymes (CYP) and transporters that cannot be held for 3 days prior to Day 1 and during treatment days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-12-17 (Actual); Primary Completion 2022-02-08 (Actual); Study Completion 2022-02-14 (Actual)

PRIMARY OUTCOMES:
Evaluation of safety and identification of the MTD/RP2D for L-Annamycin | Day 1 through Day 28
  The number of patients who experience dose-limiting toxicities (DLT) will be captured at each dose level of L-Annamycin in order to determine the MTD/RP2D

SECONDARY OUTCOMES:
Pharmacokinetics - Area under the plasma concentration | Day 1 and Day 3
  Area under the plasma concentration - time curve (AUC) of annamycin and its metabolite, annamycinol
Anti-leukemic activity | Between Day 15 and Day 35 (+/- 3 days)
  Determined by acute myeloid leukemia (AML) response rate based on the International Working Group (IWG) Response Criteria in AML (Cheson, 2003). Leukemia response rate will be evaluated by the investigator at the end of each L-Annamycin cycle based on bone marrow aspirate and peripheral blood evaluations.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Shepard, MD, Study Director — Moleculin Biotech, Inc.
Locations (5):
- Poland (5):
  - Medical University of Lodz, Lodz
  - Szpital Kliniczny Przemienienia Pańskiego Uniwersytetu Medycznego im. Karola Marcinkowskiego, Poznan
  - Samodzielny Publiczny Szpital Kliniczny nr 1 im. Prof. Tadeusza Sokołowskiego w Szczecinie, Klinika Hematologii z Oddziałem Transplantacji Szpiku, Szczecin
  - Instytut Hematologii i Transfuzjologii, Klinika Hematologii, Warsaw
  - Samodzielny Szpital Kliniczny nr 1, Wroclaw

IPD SHARING:
Plan to Share IPD: Undecided